CLINICAL TRIAL: NCT02723617
Title: The Dose-Response Effects of Lean Beef in a Mediterranean-Style Dietary Pattern on Cardiovascular Disease Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, David Baer, Supervisory Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HS54
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MED 0.5 (Other)
  Interventions: Other: MED 0.5
- MED 2.5 (Other)
  Interventions: Other: MED 2.5
- MED 5.5 (Other)
  Interventions: Other: MED 5.5
- AAD 2.5 (Other)
  Interventions: Other: AAD 2.5

INTERVENTIONS:
Other: MED 0.5 — Participants will be fed a Mediterranean diet providing 0.5 oz. per day of lean beef.
  Arms: MED 0.5
Other: MED 2.5 — Participants will be fed a Mediterranean diet providing 2.5 oz. per day of lean beef.
  Arms: MED 2.5
Other: MED 5.5 — Participants will be fed a Mediterranean diet providing 5.5 oz. per day of lean beef.
  Arms: MED 5.5
Other: AAD 2.5 — Participants will be fed an average American diet providing 2.5 oz. per day of lean beef.
  Arms: AAD 2.5

SUMMARY:
The objective of this study is to evaluate the effects of different quantities of lean beef (0.5, 2.5, 5.5 oz/day) on lipids, lipoproteins, and vascular health endpoints in the context of a modified Mediterranean dietary pattern that is representative of foods typically consumed in the United States.

DETAILED DESCRIPTION:
The DASH (Dietary Approaches to Stop Hypertension) dietary pattern, the USDA Food Pattern, and the American Heart Association (AHA) Diet are all recommended for the reduction of LDL-C and blood pressure, two major risk factors for cardiovascular disease (CVD). The recommended food-based dietary patterns emphasize consumption of vegetables, fruits and whole grains; include low-fat dairy products, poultry, fish, legumes, non-tropical vegetable oils and nuts; and limit intake of sweets, sugar-sweetened beverages and red meats. The Mediterranean dietary pattern has gained widespread popularity because of an impressive evidence base showing health benefits in the prevention of many chronic diseases including CVD. The Mediterranean Diet Pyramid recommends that red meat be consumed less than 2 servings per week, with an emphasis on lean cuts. However, as the BOLD (Beef in an Optimal Lean Diet) study has demonstrated, lean beef can be included in a heart healthy dietary pattern that achieves both low density lipoprotein and blood pressure-lowering effects. The BOLD study utilized beef consumption levels of 4 or 5.4 ounces of lean beef daily, which is significantly higher than the American average of app. 3 ounces per day. This study will evaluate three levels of beef in the context of a Mediterranean diet, compared to an Average American diet.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 20 and 40 kg/m2
* Non-smoker
* Fasting glucose ≤ 126 mg/dl

Exclusion Criteria:

* Low HDL-C (<15th percentile of US population)
* Use of cholesterol lowering medications
* Elevated blood pressure (systolic blood pressure > 160 mm Hg and diastolic blood pressure > 100 mm Hg) or use of medication to treat hypertension for less than 6 months
* Elevated triglycerides ( > 350 mg/dL)
* Active cardiovascular disease (such as a heart attack or procedure within the past six months or participation in a cardiac rehabilitation program within the last six months, stroke, or history/treatment for transient ischemic attacks in the past six months, or documented history of pulmonary embolus in the past six months)
* Presence of kidney disease, liver disease, gout, untreated or unstable hyper- or hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* Weight loss of ≥ 10% of body weight within 6 months prior to enrolling in the study
* Smokers or use of any tobacco products in past 6 months
* Known (self-reported) allergy or adverse reaction to study foods
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Lipid/lipoprotein profile will be measured in blood | Week 0, end of diet period 1 (week 4), end of diet period 2 (week 9), end of diet period 3 (week 15), end of diet period 4 (week 21)
  The following will be measured in the blood on 2 consecutive days at baseline (start of trial) and the end of each 4-week diet period: lipids and lipoproteins, apolipoproteins, lipoprotein particle number/size, and proprotein convertase subtilisin/kexin type 9 (PCSK9).

SECONDARY OUTCOMES:
Pulse Wave will be measured using Sphygmocor EXCEL | Week 0, end of diet period 1 (week 4), end of diet period 2 (week 9), end of diet period 3 (week 15), end of diet period 4 (week 21)
  Pulse wave analysis and pulse wave velocity will be conducted.
Markers of vascular health will be measured in blood | Week 0, end of diet period 1 (week 4), end of diet period 2 (week 9), end of diet period 3 (week 15), end of diet period 4 (week 21)
  Adhesion molecules and endothelin-1 will be measured in the blood.
Systemic inflammation will be measured in blood | Week 0, end of diet period 1 (week 4), end of diet period 2 (week 9), end of diet period 3 (week 15), end of diet period 4 (week 21)
  Markers of systemic inflammation will be measured, such as fibrinogen, IL-6, TNF-alpha, serum amyloid A, and CRP.
Fecal microbiota will be analyzed | Week 0, end of diet period 1 (week 4), end of diet period 2 (week 9), end of diet period 3 (week 15), end of diet period 4 (week 21)
  Feces will be analyzed for bacterial typing.
Measures of oxidative stress will be measured in urine | Week 0, end of diet period 1 (week 4), end of diet period 2 (week 9), end of diet period 3 (week 15), end of diet period 4 (week 21)
  Urinary 8-iso-PGF-2α and urinary 15-keto-dihydro- PGF-2α will be measured.
Blood glucose, serum insulin, and insulin c-peptide will be measured. | Week 0, end of diet period 1 (week 4), end of diet period 2 (week 9), end of diet period 3 (week 15), end of diet period 4 (week 21)
  Blood glucose and serum insulin and insulin c-peptide will be measured.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland
  - Penn State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DiMattia ZS, Zhao J, Hao F, Koshkin S, Bisanz JE, Patterson AD, Fleming JA, Kris-Etherton PM, Petersen KS. Effect of Varying Quantities of Lean Beef as Part of a Mediterranean-Style Dietary Pattern on Gut Microbiota and Plasma, Fecal, and Urinary Metabolites: A Randomized Crossover Controlled Feeding Trial. J Am Heart Assoc. 2025 Oct 7;14(19):e041063. doi: 10.1161/JAHA.125.041063. Epub 2025 Sep 19. PMID 40970516
- [Derived] Fleming JA, Petersen KS, Kris-Etherton PM, Baer DJ. A Mediterranean-Style Diet with Lean Beef Lowers Blood Pressure and Improves Vascular Function: Secondary Outcomes from a Randomized Crossover Trial. Curr Dev Nutr. 2025 Feb 22;9(4):104573. doi: 10.1016/j.cdnut.2025.104573. eCollection 2025 Apr. PMID 40201153
- [Derived] Fleming JA, Kris-Etherton PM, Petersen KS, Baer DJ. Effect of varying quantities of lean beef as part of a Mediterranean-style dietary pattern on lipids and lipoproteins: a randomized crossover controlled feeding trial. Am J Clin Nutr. 2021 May 8;113(5):1126-1136. doi: 10.1093/ajcn/nqaa375. PMID 33826691